CLINICAL TRIAL: NCT05527925
Title: Effects of Visual Reconstruction on Brain Function and Structure in Children With Congenital Cataract
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Professor, Sun Yat-sen University
Other Study IDs: 2019KYPJ055
Record Dates: First submitted 2022-08-30; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Congenital Cataracts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Congenital cataracts children (0~3 years): Children with congenital cataracts between the ages of 0 and 3 years
  Interventions: Device: MRI
- Normal children (0~3 years): Children without congenital cataracts between the ages of 0 and 3 years
  Interventions: Device: MRI
- Congenital cataracts children (6~18 years): Children with congenital cataracts between the ages of 6 and 18 years
  Interventions: Device: MRI
- Normal children (6~18 years): Children without congenital cataracts between the ages of 6 and 18 years
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — Brain testing of patients using MRI

SUMMARY:
Children have considerable plasticity of the visual system during the formation and maturation of various visual functions at different ages. Congenital cataracts are the leading cause of treatable blindness in children. With the continuous improvement of surgical approaches and surgical techniques, the success rate of congenital cataract surgery has been significantly improved clinically, and the visual function of children has been significantly improved after surgery. However, to date, there has been no experimental study of specific changes in the brain before and after surgery in children with congenital cataracts to explore its relationship with visual reconstruction. We aim to investigate the effects of congenital cataract surgery on the brain function and structure of children through preoperative and postoperative analysis and comparison of brain imaging such as BOLD-fMRI and DTI, and provide new ideas for the clinical treatment and prognostic assessment of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Children with congenital cataracts

Exclusion Criteria:

* Other oculo-cerebral and systemic diseases that may affect the outcome

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with congenital cataracts
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from functional magnetic resonance imaging | 1 week before surgery , 1 month, 3 month, 6 month after surgery

SECONDARY OUTCOMES:
Change from best corrected visual acuity | 1 week before surgery , 1 month, 3 month, 6 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, Study Director — Study Principal Investigator
Locations (1):
- SunYat-senU, Guangzhou, Guangdong, China